CLINICAL TRIAL: NCT06530329
Title: Investigation of the Short-Term Effects of Ischemic Compression Applied in Addition to Classical Massage on Pain, Functionality and Quality of Life in the Treatment of Myofascial Trigger Points on the Upper Trapezius Muscle in Women
Brief Title: Short-Term Effects of Ischemic Compression Applied in Addition to Classical Massage in the Treatment of Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, PT, MSc., Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28.07.2024-EDP&DA
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Classical massage group
  Interventions: Other: Classical massage
- Group 2 (Experimental): Classical massage + ischemic compression group
  Interventions: Other: Classical massage; Other: Ischemic compression

INTERVENTIONS:
Other: Classical massage — Classical massage was started by general stroking 3 times. Then, it was continued by kneading 3 times. After the kneading movement, fibrocytic nodules on the muscle were searched and friction was applied to the found nodules one by one. The massage of the muscle was completed by applying stroking 3 times. The application was carried out 3 times a week for 2 weeks to evaluate the short-term effect.
Other: Ischemic compression — Ischemic compression was applied to the trigger points in the upper trapezius muscle using an average pressure of 1 kg at a right angle, and after compression, passive stretching was applied to the upper trapezius muscle 3 times in 20-second periods. The application was performed 3 times a week for 2 weeks to evaluate the short-term effect.
  Arms: Group 2

SUMMARY:
The aim of our study was to investigate the short-term effects of ischemic compression applied in addition to classical massage for the treatment of myofascial trigger points on the upper trapezius muscle in women on pain, functionality and quality of life.

DETAILED DESCRIPTION:
The aim of our study was to investigate the short-term effects of ischemic compression applied in addition to classical massage in the treatment of myofascial trigger points on the upper trapezius muscle in women on pain, functionality and quality of life. "Visual Analog Scale (VAS)" was used for pain assessment of individuals who accepted to participate in the study; universal goniometer was used to measure active neck active range of motions (AROM) for functionality; and "Short Form-36 (SF-36)" was used for quality of life. Then, the participants were randomly divided into two groups [Group 1: classical massage group; Group 2: classical massage + ischemic compression group]. Classical massage was applied to both groups three times a week for two weeks, and ischemic compression was applied to Group 2 in addition to classical massage. At the end of the treatment period, the participants were re-evaluated in terms of VAS, neck AROM and SF-36 scores.Statistical analysis will be performed with SPSS 24.0 program. If the data is parametric, paired sample t-test will be used for within-group evaluation; independent sample t-test will be used for between-group evaluation. If the data is non-parametric, Wilson test will be used for within-group evaluation and Mann Whitney U test will be used for between-group evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-50
* Having a myofascial trigger point detected in the upper trapezius muscle for at least two weeks
* Being a student or staff of Halic University
* Being literate

Exclusion Criteria:

* Having a history of cervical surgery
* Having a malignant disease
* Pregnancy
* Menopause
* Having cooperation problems

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female
Enrollment: 22 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | at baseline and at week 2.
  Pain assessment was made with Visual Analog Scale (VAS). The subjects were informed that the number '0' on a 10 cm horizontal line indicated 'no pain' and the number '10' indicated 'unbearable pain'. The subjects were asked to mark the pain they felt on the VAS scale for 3 different areas, namely trapezius pain, neck pain and headache, and the points they marked were recorded as the severity of pain in cm. VAS measurements were performed twice in total, before and after treatment.
Active Range of Motion | at baseline and at week 2.
  Active Range of Motion (AROM) measurement was evaluated using a universal goniometer. While the patient was in a sitting position, the pivot point, fixed arm and movable arm of the goniometer were placed in the specified reference areas. The patient was asked to actively perform neck flexion, extension, right-left lateral flexion and right-left rotation movements and the values at the end of the movements were recorded in degrees. AROM measurements were performed twice in total, before and after treatment.
Short-Form 36 | at baseline and at week 2.
  The Short Form-36 (SF-36) scale was used to assess quality of life. The lowest score represents the worst health status. SF-36 measurement was performed twice, before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Sahin Altac, PT, MSc., Principal Investigator — Halic Üniversity
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683
- [Result] Bethers AH, Swanson DC, Sponbeck JK, Mitchell UH, Draper DO, Feland JB, Johnson AW. Positional release therapy and therapeutic massage reduce muscle trigger and tender points. J Bodyw Mov Ther. 2021 Oct;28:264-270. doi: 10.1016/j.jbmt.2021.07.005. Epub 2021 Jul 14. PMID 34776151
- [Result] Cagnie B, Castelein B, Pollie F, Steelant L, Verhoeyen H, Cools A. Evidence for the Use of Ischemic Compression and Dry Needling in the Management of Trigger Points of the Upper Trapezius in Patients with Neck Pain: A Systematic Review. Am J Phys Med Rehabil. 2015 Jul;94(7):573-83. doi: 10.1097/PHM.0000000000000266. PMID 25768071
- [Result] Sahin D, Kaya Mutlu E, Sakar O, Ates G, Inan S, Taskiran H. The effect of the ischaemic compression technique on pain and functionality in temporomandibular disorders: A randomised clinical trial. J Oral Rehabil. 2021 May;48(5):531-541. doi: 10.1111/joor.13145. Epub 2021 Jan 21. PMID 33411952